CLINICAL TRIAL: NCT00185874
Title: A Phase I Trial of Intratumoral Dendritic Cell Immunotherapy in Thermally Ablated Liver Metastases
Brief Title: Phase I Intratumoral Dendritic Cell Immunotherapy in Thermally Ablated Liver Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to lack of funding
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Edgar G Engleman, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP0002; HEP0002; NCT00185874; NIH 16766
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

INTERVENTIONS:
Biological: Intratumoral Dendritic Cell Immunotherapy
Biological: autologous dendritic cells

SUMMARY:
Up to twenty-two patients will be enrolled in this study to receive autologous dendritic cells (DCs) administered intratumorally into liver metastases following radiofrequency thermal ablation of those lesions. Patients will receive two vaccinations of DCs at monthly intervals. A dose escalation study of DCs will be included in this study in an attempt to define the maximum tolerated dose of administered DCs.

ELIGIBILITY:
Inclusion Criteria:- Patients must have a histologically confirmed colorectal or neuroendocrine cancer with two or more hepatic metastatic lesions.

* Patients must have unresectable liver metastasis by virtue of:

  * Bi-lobar disease.
  * Extra-hepatic disease.
  * Patients for whom there are medical contraindications to surgery.
  * Anatomic sites within the liver that in the opinion of our surgeon would likely be left with positive margin.
* Patient must have a minimum of 2 RFA-eligible lesion in the liver. Such as hepatic lesions that are 5 cm or smaller and that are accessible to RF ablation, which in general excludes sites contiguous with critical structures such as bowel or central bile duct and also those that are not amenable to radiographic localization such as small lesions in the dome of the liver. Extra-hepatic disease will be allowed provided that the liver lesions represent the most life-threatening site for that patient. Examples include sub centimeter asymptomatic lung metastases or asymptomatic retroperitoneal lymph nodes or peritoneal metastases
* Evaluable disease by CT scan or MRI in addition to the lesions to be treated with RFA.
* More than 4 weeks must have elapsed from the time of major surgery or completion of the last dose of chemotherapy, radiation therapy, investigational therapy and patients must adequately recover from these effects.
* Life expectancy of >3 months.
* Karnofsky performance status >70%.
* Patients must have normal organ and marrow functions as defined below:

  * absolute neutrophil count >1,500/mm^3
  * platelets >70,000/mm^3
  * total bilirubin <1.5 mg/dL
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >60mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
  * albumin > 2.8 mg/dL
* Patients must have adequate clotting function (platelet > 70k; INR<1.4; PTT<60).
* Age >18 years.
* The effects of DCs on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* No history of autoimmune diseases.
* Ability to understand the willingness to sign a written informed consent document. Exclusion Criteria:- Patients may not be receiving anticoagulation therapy.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases will be excluded because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse effects.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Patients with a history of portal hypertension, cirrhosis/hepatitis, or with radiographic evidence of cirrhosis and/or varices are at high risk for developing a complication when undergoing a liver biopsy and may be excluded at the investigators' discretion from participation in this protocol.
* Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of harvesting autologous dendritic cells (DC) for CT-guided intratumoral DC injection | NA- study terminated
To establish the maximally tolerated dose (MTD) and dose limiting toxicity (DLT) of intratumoral autologous dendritic cell vaccination in combination with radiofrequency ablation (RFA) of liver metastases. | NA- study terminated
To determine the toxicity of this regimen | NA- study terminated

SECONDARY OUTCOMES:
To determine the activity of this regimen as determined by tumor marker response, pathologic response and radiographic response of treated lesions. | NA- study terminated
To evaluate the immune response of patients treated with RFA + DC based on the presence and characterization of tumor infiltrating white blood cells | NA- study terminated

CONTACTS AND LOCATIONS:
Overall Officials: Edgar G Engleman, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States